CLINICAL TRIAL: NCT07066215
Title: Effects of Range of Motion, Balance and Muscle Strength on Functional Capacity in Knee Osteoarthritis
Brief Title: Effects of Range of Motion, Balance and Muscle Strength in Knee Osteoarthritis
Status: Recruiting | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Kübra Alpay, Lecturer of Physiotherapy and Rehabilitation Department, Bezmialem Vakif University
Other Study IDs: KA25-1
Record Dates: First submitted 2025-07-14; First posted 2025-07-15 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Primary Knee Osteoarthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Knee osteoarthritis (OA) is a chronic and progressive joint disease characterized by the degeneration of articular cartilage, subchondral bone sclerosis, and the formation of osteophytes. This condition leads to joint pain and stiffness, negatively affecting individuals' quality of life. Joint stiffness, decreased quadriceps strength, and impaired proprioceptive sensation result in functional limitations. Due to these symptoms, individuals experience difficulties in performing daily activities such as rising from a chair, walking, and climbing stairs. The aim of this study is to evaluate the effects of joint range of motion, balance, and muscle strength on functional capacity in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
In knee OA, structural changes in the cartilage and the formation of peripheral osteophytes contribute to joint stiffness and a reduction in the range of motion, which adversely affects physical function, particularly in older adults. Activities such as stair climbing, sitting and standing, and walking require the contribution of core muscles as well as lower extremity muscles, particularly the knee extensors. In knee OA, there is a reported decrease in lower extremity muscle strength, especially in the quadriceps femoris muscle, which further impairs functional activities in the advanced stages of the disease.

Arthritic damage to joint mechanoreceptors in osteoarthritis leads to a decline in motor control and proprioceptive sensitivity. These sensorimotor deficits result in decreased stability and impaired balance function. Additionally, reduced muscle strength can hinder neuromuscular control, leading to postural instability and an increased risk of falls, especially in older patients.

Identifying the factors that contribute to the decline in functional capacity is crucial for planning appropriate exercise programs. The aim of this study is to evaluate the effects of joint range of motion, balance, and muscle strength on functional capacity in patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Primary knee osteoarthritis

Exclusion Criteria:

* Previous surgery in the lower extremity
* Neuromuscular disease
* Vestibular pathology
* Physiotherapy intervention or intra-articular injection within the last 6 months

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have diagnosed primary knee osteoarthritis will be included
Sampling Method: Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Range of motion | Baseline
  Knee flexion range of motion measurement with goniometer
Muscle strength | Baseline
  Muscles strength measurement with hand-held dynamometer for knee extensor muscle
Balance | Baseline
  Biodex Balance System will be used for postural stability evaluation. Lower scores indicate better stability and higher scores mean poor balance.
6-minute walk test | Baseline
  Walking distance will be measured
5 time sit-to-stand test | Baseline
  Test completion time will be evaluated
Stair climb test | Baseline
  Test completion time will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Kubra Alpay, PhD, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Eyup, Turkey (Türkiye)